CLINICAL TRIAL: NCT06445751
Title: Step up for STEM and Health Careers: An Interactive Digital Resource to Reduce STEM-related Biases and Improve High School STEM Learning Environments
Brief Title: Step Up for STEM and Health Careers
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Funding was terminated pursuant to the Fiscal Year 2003 National institutes of Health ("NIH") Grants Policy Statement, and 2 C.F.R. 200.340(a)(2).
Sponsor: Ohio State University (Other)
Collaborators: Resilient Games Studio (Industry); University of Chicago (Other); National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Nicole Thomas, Research Scientist, CATALYST, Ohio State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2023B0273
Record Dates: First submitted 2024-05-21; First posted 2024-06-06 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2024-05

CONDITIONS: Adolescent Behavior
Keywords: STEM; Adolescents; Diversity; Digital Games
MeSH Terms: conditions — Adolescent Behavior | interventions — Microscopy, Electron, Scanning Transmission; Health Personnel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Step Up for STEM Careers Game Intervention (Experimental): Youth in the intervention group will play a six-episode, interactive game on the importance of diversity in STEM and health careers, STEM/health career self-efficacy, and creating an inclusive learning environment for others. This includes featuring diverse youth who model STEM/health self-efficacy; integrating STEM/health professional characters as "in-game" content experts and role models; and incorporating mini games to reinforce skills and behavior.
  Interventions: Behavioral: Step Up for STEM and Health Careers ("Step Up") game
- Educational PowerPoint (Active Comparator): Youth in the comparator group will complete an educational PowerPoint presentation on the importance of diversity in STEM and health careers, STEM/health career self-efficacy, and creating an inclusive learning environment for others. This PowerPoint presentation will contain sections that correspond to each episode of the Step Up for STEM and Health Careers intervention.
  Interventions: Behavioral: Educational PowerPoint Presentation on Diversity in STEM Careers

INTERVENTIONS:
Behavioral: Step Up for STEM and Health Careers ("Step Up") game — Step Up for STEM and Health Careers ("Step Up") game is an interactive, digital resource to help high school students understand the importance of diversity in STEM and health careers, attain STEM/health career self-efficacy, and help them create an inclusive learning environment for others.
  Arms: Step Up for STEM Careers Game Intervention
Behavioral: Educational PowerPoint Presentation on Diversity in STEM Careers — An educational PowerPoint on Diversity in STEM careers to increase adolescents' STEM/health career self-efficacy, and help them create an inclusive learning environment for others.
  Arms: Educational PowerPoint

SUMMARY:
The goal of this randomized controlled trial is to evaluate "Step Up for STEM and Health Careers". The "Step Up for STEM and Health Careers" ("Step Up") game is an interactive, digital resource that includes the key elements of a bystander intervention for high school students to understand the importance of diversity in STEM; it also addresses skills, attitudes, and awareness to attain positive STEM identities and mitigate bias and harassment in STEM and health learning environments.

Participants in the intervention arm will be asked to complete the Step Up interactive game; participants in the comparison group will be asked to view a PowerPoint presentation on bias and harassment in STEM/health fields as the control experience. The Step Up game intervention and study outcomes are theory-based (Theory of Planned Behavior, Social Cognitive Career Theory (SCCT)): we will assess the impact of Step Up on attitudes about STEM/health careers, STEM/health career self-efficacy, and bystander behavior.

DETAILED DESCRIPTION:
The goal of this randomized control trial is to evaluate the impact of the "Step Up for STEM and Health Careers" intervention game on STEM/health career and bystander attitudes, as well as self-efficacy. Participants will be randomly assigned to participate in either the Step Up intervention game or the educational PowerPoint presentation.

The "Step Up for STEM and Health Careers" intervention consists of students playing a "Step Up" game to help them understand the importance of diversity in STEM and health careers, attain STEM/health career self-efficacy, and create an inclusive learning environment for others. The control group consists of an educational PowerPoint presentation on the importance of diversity in STEM and health careers, STEM/health career self-efficacy, and creating an inclusive learning environment for others.

The Step Up intervention game (created by Resilient Games Studio (RGS)) consists of six digital episodes that focus on a specific topic: importance of diversity in STEM careers, heuristics and biases, structural biases and intersectionality, harassment, sexual harassment, and bystander behaviors. Each episode includes interactive mini-games to teach theory-based skills and lessons. Adult characters, who serve as "in-game" STEM/health role models, are integrated throughout the game. The game was built based on the Theory of Planned Behavior (TPB) and the Social Cognitive Career Theory (SCCT) to improve STEM/health career and bystander attitudes, as well as self-efficacy.

The educational PowerPoint presentation on bias and harassment in STEM/health fields was also created by RGS and will be used as a control experience for adolescent participants. The PowerPoint presentation will contain sections that correspond to each of the episode topics of the Step Up intervention game.

ELIGIBILITY:
Inclusion Criteria:

* English-speaking
* Access to a computer and internet connection
* Live in Chicago Metropolitan Area
* Current high school student (enrolled in grade 9-12); or in 12th grade in 2023-2024 school year

Exclusion Criteria:

-

Ages: 13 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 24 (Actual)
Dates: Start 2024-07-02 (Actual); Primary Completion 2025-03-21 (Actual); Study Completion 2025-03-21 (Actual)

PRIMARY OUTCOMES:
STEM/health career attitudes using modified Career Interest (Christensen, et al., 2014) and STEM Semantics (Knezek and Christensen, 2008) questionnaires | From baseline pre-test immediately preceding randomization to post-test up to 3 days post intervention/comparator
  One's beliefs about outcomes associated with STEM/health careers
STEM/health career self-efficacy using a modified Career Interest Questionnaire (Christensen, et al., 2014) | From baseline pre-test immediately preceding randomization to post-test up to 3 days post intervention/comparator
  The perception one has the requisite skills and capabilities for attaining a STEM/health career

SECONDARY OUTCOMES:
Intent to pursue a STEM/health career using a modified Career Interest Questionnaire (Christensen, et al., 2014) | From baseline pre-test immediately preceding randomization to post-test up to 3 days post intervention/comparator
  One's intent to pursue a STEM/health career
Knowledge of the value of diversity in STEM/health careers using a questionnaire | From baseline pre-test immediately preceding randomization to post-test up to 3 days post intervention/comparator
  One's knowledge of the value of diversity in STEM/health careers
Intent to intervene as a bystander when witnessing harassment on the basis of race, gender, disability status, etc., using a questionnaire derived from the Bystander Questionnaire (Garza et al., 2023; McMahon and Banyard, 2012) | From baseline pre-test immediately preceding randomization to post-test up to 3 days post intervention/comparator
  One's intent to intervene as a bystander when witnessing harassment on the basis of race, gender, disability status, etc.

CONTACTS AND LOCATIONS:
Overall Officials: Tim Parsons, Study Director — Resilient Games Studio
Locations (1):
- Ohio State University, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No